CLINICAL TRIAL: NCT07308847
Title: Horizon 360 Protocol for the Treatment of Paroxysmal Atrial Fibrillation With the Prospective, Single Arm, Unblinded Pre-market Clinical Study to Evaluate the Safety and Effectiveness of the Sphere-360 Catheter and Affera Mapping and Ablation System for Treating Paroxysmal Atrial Fibrillation (PAF)
Brief Title: Horizon 360 Protocol for the Treatment of Paroxysmal Atrial Fibrillation With the Sphere-360™ Catheter and Affera™ Mapping and Ablation System (Horizon 360)
Acronym: Horizon 360
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Ablation Solutions (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Horizon 360
Record Dates: First submitted 2025-12-26; First posted 2025-12-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal AF
Keywords: Paroxysmal Atrial Fibrillation; Atrial Fibrillation; Pulsed Field Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Pulmonary Vein Isolation Ablation (Experimental): Pulmonary Vein Isolation Ablation utilizing the Sphere-360 and Affera Mapping and Ablation System
  Interventions: Device: Sphere-360 Pulsed Field Ablation Catheter with the Affera Mapping and Ablation System

INTERVENTIONS:
Device: Sphere-360 Pulsed Field Ablation Catheter with the Affera Mapping and Ablation System — Pulmonary Vein Isolation using the Sphere-360 Pulsed Field Ablation Catheter with the Affera Mapping and Ablation System

SUMMARY:
The study is a prospective, single-arm, pre-market clinical study and will enroll up to 300 subjects at up to 26 sites in the United States (US) for analysis of primary objectives. No single site may contribute more than 15% of the enrollments.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of recurrent symptomatic PAF, which is defined as continuous AF episode lasting longer than 30 seconds but terminates spontaneously or with intervention within 7 days of onset, documented by the following:

   1. a physician's note indicating at least 2 symptomatic PAF episodes occurring within 6 months prior to enrollment; and
   2. at least 1 electrocardiographically documented episode within 12 months prior to enrollment
2. Adults who are ≥18 and ≤80 years of age on the day of enrollment.
3. Willing and able to comply with all baseline and follow-up evaluations for the full length of the study.

Exclusion Criteria:

1. Continuous AF lasting more than 7 days. This includes persistent atrial fibrillation (PsAF) (both early or long-standing) by diagnosis or continuous duration > 7 days
2. AF that required three (3) or more distinct cardioversions in the preceding 12 months.
3. LA anteroposterior > 5.0 cm (by MRI, CT, or TTE)
4. Any of the following procedures, implants, or conditions at baseline: prior left atrial catheter or surgical ablation, prior left atrial percutaneous interventions including left atrial appendage occlusion, and septal closure devices
5. Planned LAA closure procedure or implant of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function) for any time during the follow-up period
6. Patient who is not on oral anticoagulation therapy for at least 3 weeks prior to the ablation procedure
7. Presence of a permanent pacemaker, biventricular pacemaker, loop recorder/insertable cardiac monitor (ICM), or any type of implantable cardiac defibrillator (with or without biventricular pacing function)
8. Presence of any pulmonary vein stents
9. Known pre-existing pulmonary vein stenosis
10. Pre-existing hemidiaphragmatic paralysis
11. Prior valvular (surgical or percutaneous) procedure including prosthetic, bioprosthetic, valve replacement, valve repair or valvuloplasty, and any prior atriotomy
12. Moderate to severe aortic or mitral valve stenosis
13. Moderate to severe mitral regurgitation (i.e., 3+ or 4+ MR)
14. Any cardiac surgery, myocardial infarction, PCI / PTCA or coronary artery stenting which occurred during the 3-month interval preceding the consent date
15. Unstable angina
16. NYHA Class III or IV congestive heart failure or documented left ventricular ejection fraction (LVEF) less than or equal to 40% measure by acceptable cardiac testing (e.g. TTE), or planned transplant or left ventricular assist device (LVAD)
17. Severe lung disease, primary pulmonary hypertension, or any lung disease with abnormal blood gases or requiring supplemental oxygen
18. Rheumatic heart disease
19. Severe thrombocytosis, thrombocytopenia, or any bleeding or clotting disorder
20. Contraindication to or unwillingness to use systemic anticoagulation
21. Documented left atrial thrombus on imaging
22. Active systemic infection or sepsis
23. Hypertrophic cardiomyopathy
24. Known reversible causes of AF, including but not limited to uncontrolled hyperthyroidism, severe untreated obstructive sleep apnea, and acute alcohol toxicity
25. Any cerebral ischemic event (strokes or TIAs) which occurred during the 6-month interval preceding the consent date
26. Carotid stenting or endarterectomy
27. History of thromboembolic event within the past 6 months or evidence of intracardiac thrombus at the time of the procedure
28. Any woman known to be pregnant or breastfeeding, or any woman of childbearing potential who is not on a reliable form of birth regulation method or abstinence
29. Patient with life expectancy that makes it unlikely 12 months of follow-up will be completed
30. Current or anticipated participation in any other clinical trial of a drug, device or biologic during the duration of the study not pre-approved by Medtronic
31. Known allergies or hypersensitivities to adhesives
32. Body mass index > 40 kg/m2
33. Atrial myxoma
34. Significant restrictive or obstructive pulmonary disease or chronic respiratory condition.
35. Renal insufficiency with an estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2, or any history of renal failure requiring dialysis or renal transplant
36. Solid organ or hematologic transplant, or currently being evaluated for an organ transplant
37. Presence of intramural thrombus, tumor, or other abnormality that precludes vascular access, catheter introduction, or manipulation
38. Known drug or alcohol dependency
39. Significant congenital anomaly or medical problem that, in the opinion of the investigator, would preclude enrollment in this study or compliance with follow-up requirements or would impact the scientific soundness of the clinical trial results.
40. Treatment with Amiodarone within the 3 months prior to enrollment
41. Amyloid heart disease (cardiac amyloidosis)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2027-11-22 (Estimated); Study Completion 2027-11-22 (Estimated)

PRIMARY OUTCOMES:
Freedom from Atrial Tachyarrhythmia Recurrence Through 12 Months Post-Ablation | Index ablation procedure through 12 months of follow up.
  Freedom from documented recurrence of atrial fibrillation, atrial tachycardia, or atrial flutter based on electrocardiographic data through 12 months (365 days) and excluding a 90-day blanking period. The study requires 24-hour Holter monitoring at 6 and 12 months in addition to weekly and symptomatic trans-telephonic monitoring (TTM) transmissions through 12 months, and 12-lead ECGs at all follow up visits. Atrial tachyarrhythmia observed via any of those instruments, as well as acute procedural failure, repeat ablation, cardioversion, an increase in anti-arrhythmic drugs, or use of amiodarone at any time during the study will constitute a failure.
Incidence of Device- and Procedure-Related Serious Adverse Events Through 6 Months | Index ablation procedure through 6 months of follow up.
  Primary safety events (device- and procedure-related serious adverse events, as adjudicated by the Clinical Events Committee) for the Sphere-360 Catheter and Affera Mapping and Ablation System:
  Within 7 days: heart block, major bleeding needing transfusion, MI, permanent phrenic nerve paralysis, pulmonary edema, severe pericarditis, significant effusion/tamponade, stroke/CVA, systemic/pulmonary embolism needing intervention, TIA, vagal nerve injury causing esophageal dysmotility/gastroparesis, vascular access complications needing intervention, AKI needing dialysis or hospitalization >48h or prolonged >48h, death, any device/procedure-related CV/pulmonary event causing/prolonging hospitalization >48h (excludes recurrent AF/AT/AFL).
  Within 3 months: atrioesophageal/esophago-pericardial fistula, esophageal perforation (device/procedure related; excludes TEE/nasogastric tube injury).
  Within 6 months: pulmonary vein stenosis (≥70% diameter reduction).

SECONDARY OUTCOMES:
Secondary Endpoint: Quality of Life (AFEQT) | Index ablation procedure through 12 months of follow up.
  Change in AFEQT score from baseline to 12 months. The AFEQT is an AF-specific health-related quality of life questionnaire, scored 0-100 (higher scores indicate better quality of life).
Secondary Endpoint: Quality of Life (EQ-5D) | Index ablation procedure through 12 months follow up.
  Change in EQ-5D composite score from baseline to 12 months. The EQ-5D is a standardized instrument for generic health status, with composite scores indexed to a US reference population.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Reddy, MD, Principal Investigator — Icahn School of Medicine at Mt Sinai
Locations (4):
- United States (4):
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Southcoast Health System, Fall River, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Northwell Health Lenox Hill Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No